CLINICAL TRIAL: NCT05708417
Title: A Weight-Neutral Approach for a Healthier Lifestyle Among Obesity - A Lifestyle Intervention Anchored in The South Danish Obesity Initiative (SDOI).
Brief Title: A Weight-Neutral Approach for a Healthier Lifestyle Among Obesity - A Lifestyle Intervention Anchored in SDOI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Lifestyle_intervention_SDOI
Record Dates: First submitted 2023-01-13; First posted 2023-02-01 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Health Related Quality of Life and Weight Condition

STUDY DESIGN:
Intervention Model Description: The study is a one-site, single-blind, clinical intervention study.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight neutral intervention (Experimental): The intervention is based on the concept of Acceptance and Commitment Therapy (ACT) and is conducted by specially trained physiotherapist and a dietician. The intervention in SDOI has the predominantly focus on each individual reflection and realization and is built upon ACT' six core processes. Specific focus on teach participant with different narrative and background and on coaching and back-and-forth dialogue with physiotherapist and dietician. The program is based on up to 13 times attendance within the 12 months intervention period. Part 1: Three to five individual coaching, Part 2: six group sessions and Part 3: one or two individual coaching.
  Compliance to the intervention is classified as 'good' if the participants participate for a minimum four out of six group sessions, a minimum three out of five initial individual coaching and a minimum one out of two individual coaching post intervention.
  Interventions: Behavioral: Lifestyle Intervention
- Reference group (Placebo Comparator): The reference group will not receive the intervention in the study and only participate in the test/data collection. The reference group will established consisting of participants participating in the SDOI program but, who of some reasons have refused participating in the lifestyle program. In case of insufficient recruitment of participants to the reference group, individuals meeting inclusion criteria such as age and BMI will be recruited via advertising in local newspapers and social media.
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: Lifestyle Intervention — The intervention in SDOI has the predominantly focus on each individual reflection and realisation and is built upon ACT' six core processes: 1) Acceptance, 2) Cognitive defusion 3) Being present, 4) Self as context, 5) Values, and 6) Committed action.
  The program is based on up to 13 times attendance within the 12 months intervention period.
  Arms: Weight neutral intervention
Other: Placebo — No lifestyle intervention within the study, only test/datacollection
  Arms: Reference group

SUMMARY:
The study aim is to evaluate a patient-centred intervention focusing on improved quality of life and wellbeing among individuals with obesity and risk factors for adverse outcome.

DETAILED DESCRIPTION:
In Denmark, University Hospital of Southern Denmark in Esbjerg has initiated The South Danish Obesity Initiative (SDOI) to optimize the treatment of and the research in obesity. The hospital has for years, offered treatment to individuals with obesity, however, SDOI is an investigation program with the aim to identify people with undiagnosed obesity-related diseases by a systematic and stepwise approach, delivering an up-to-date treatment of diagnosed diseases and offering personalized lifestyle advice based on the finding in the investigation program. The SDOI program comprises collaboration between different medical departments at the hospital and furthermore, entails the establishment of a well-defined cohort as a basis for research. ACT is of interest in the construction of the personalized lifestyle advice in the SDOI program. However, there is limited research available on the effect of the behaviour therapy ACT as a basic method for a lifestyle program targeting overweight individuals who have been made aware of obesity related diseases and re-conditions. ACT might be a valuable tool to assist these individuals to increase their quality of life and thereby, ability to make lifestyle changes.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be eligible for inclusion if they are ≥18 years
* Body mass index above 30 kg/m2

Exclusion Criteria:

* Individuals referred for bariatric surgery will not be eligible for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
HRQoL . | 52 weeks
  Measured by the questionnaire Impact of Weight on Quality of Life-Lite at week 52. Scores range from 0 to 100, with 100 representing the best quality of life.

SECONDARY OUTCOMES:
General physical activity | 52 weeks
  Measured by Accelerometer
Body perception | 52 weeks
  Questionnaire
Isometric muscle strength | 52 weeks
  Measured by Biodex dynanometer
Self-esteem | 52 weeks
  Measured by questionnaire
Total cholesterol (mml/L) | 52 weeks
  Blood sample
Insulin resistance (HOMA-IR) | 52 weeks
  Blood sample
Diastolic and systolic Blood pressure (mm Hg) | 52 weeks
  Blood pressure monitor
Perceived chronic pain | 52 weeks
  Measured on VAS scale. The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100
Aerobic capacity | 52 weeks
  One-point Åstrand test

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bogh Juhl, Professor, Study Director — Hospital of South West Jutland, 6700 Esbjerg , Denmark
Locations (1):
- Hospital of Southwest Denmark, Esbjerg, Region Syddanmark, Denmark